CLINICAL TRIAL: NCT05790252
Title: Using the Transdermal Patch for BupRenorphine Induction DurinG PrEgnancy: A Randomized Controlled Trial (The Patch BRIDGE Trial)
Brief Title: Transdermal Patch for BupRenorphine Induction DurinG PrEgnancy (Patch BRIDGE)
Acronym: Patch BRIDGE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jeannie Kelly, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202209093
Record Dates: First submitted 2023-03-13; First posted 2023-03-30 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Pregnancy Related; Pregnancy, High Risk; Pregnancy Complications; Buprenorphine Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders; Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bridge Induction Arm (Experimental)
  Interventions: Drug: Buprenorphine Transdermal Matrix Patch
- Standard Arm (Placebo Comparator)
  Interventions: Other: Sham patch

INTERVENTIONS:
Drug: Buprenorphine Transdermal Matrix Patch — Buprenorphine transdermal patches will be applied at time of induction initiation and removed at 48 hours.
  Arms: Bridge Induction Arm
Other: Sham patch — Bandage applied at time of induction initiation and removed at 48 hours.
  Arms: Standard Arm

SUMMARY:
The goal of this clinical trial is to compare buprenorphine patch for induction (starting) of buprenorphine in pregnant patients with opioid use disorder. The main questions it aims to answer are:

1. Is there a buprenorphine induction method that results in the least moderate-to-severe opioid withdrawal symptoms in pregnant patients with opioid use disorder?
2. Is there a buprenorphine induction method that results in a higher treatment success rate? Under normal circumstances, patients who are planning to start sublingual (under the tongue) buprenorphine for opioid use disorder must first go into withdrawal to start the medication safely. Study participants will be given a buprenorphine patch during the required withdrawal period before starting sublingual treatment, and be surveyed daily by phone to assess their withdrawal symptoms. They will also be followed at prenatal appointments to evaluate treatment success based on urine drug screen results. Researchers will compare patients receiving no buprenorphine patch according to the current standard care protocol.

ELIGIBILITY:
Inclusion Criteria:

* Viable pregnancy
* Meet diagnostic criteria for opioid use disorder
* Receive prenatal care through opioid use disorder specific clinic at our institution
* Opioid use within 24 hours prior to presentation
* Desire treatment with buprenorphine

Exclusion Criteria:

* Patients already receiving treatment for opioid use disorder
* History of prior induction attempt with buprenorphine
* Active withdrawal at time of presentation
* Medical contraindication to buprenorphine
* Requiring immediate hospitalization

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Induction withdrawal severity | Days 0 through 4
  Subjective Opioid Withdrawal Scale (SOWS) scores collected during buprenorphine induction. SOWS scores range from 0-64 with higher scores representing worse withdrawal. Mild withdrawal is defined as scores 0-10, moderate as 11-20, and severe as 21+.

SECONDARY OUTCOMES:
Induction success | Days 0 through 7
  Induction success, a binary defined by fulling all of the following:
  * attendance at 1 week follow up (yes/no)
  * buprenorphine in urine at initial follow up (positive/negative on urine drug screening)
  * and absence of precipitated withdrawal (yes/no)
Treatment adherence | Days 0 through delivery
  defined as percent of urine drug screens positive for buprenorphine throughout pregnancy
Recovery success | Days 0 through delivery
  defined as percent of urine drug screens negative for non-prescribed opioids during prenatal care

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie C Kelly, MD, MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No